CLINICAL TRIAL: NCT03490422
Title: Pulpotomy in Carious Permanent Mature Teeth: Pulp Survival and Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Dr Victoria Yu, Associate Professor, National University Health System, Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-221-000-060-112
Record Dates: First submitted 2018-03-26; First posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-03

CONDITIONS: Pulpitis; Pulp Exposure, Dental; Pulp and Periapical Tissue Disease
Keywords: pulpotomy; permanent teeth; deep caries management; risk factors; clinical indicators for pulpotomy
MeSH Terms: conditions — Pulpitis; Dental Pulp Exposure | interventions — Pulpotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulpotomy (Experimental): Pulpotomy is performed in carious-exposed pulp in mature permanent teeth
  Interventions: Procedure: Pulpotomy

INTERVENTIONS:
Procedure: Pulpotomy — Pulpotomy in mature carious permanent teeth

SUMMARY:
This Trial evaluated the extent of pulp survival following pulpotomy in the permanent tooth pulp exposed by caries and identify potential risk factors for pulpal complications.

DETAILED DESCRIPTION:
Healthy patients ≥ 21 years old were recruited with informed consent. Inclusion criteria were symptomatic and asymptomatic periodontally sound teeth, positive response to pulp sensibility tests, pulp exposure by caries with bleeding, haemostasis achieved within 10 minutes and normal apical tissues. Under local anaesthesia and rubber dam isolation, caries was removed before pulpotomy. Pain complaint, clinical and radiographic data were collected during recalls for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

Patient factors:

* Male and female at least 21 years of age
* Healthy and ambulant
* Mild diseases only and without substantive functional limitations
* Able to return for scheduled recalls

Tooth factors:

* Deep caries leading to pulp exposure
* With or without pre-operative spontaneous and/or aggravated pain
* Positive response to Cold and Electric Pulp Tests
* Positive bleeding on pulp exposure
* Haemostasis within 10 minutes
* Intact and continuous periodontal ligament space and dental lamina dura on radiograph

Exclusion Criteria:

Patient factors:

* Younger than 21 years of age
* Pregnant female
* Poorly controlled systemic diseases e.g. diabetes mellitus, hypertension

Tooth factors:

* Extensive tooth structure loss requiring post and core retained restoration
* Uncontrolled periodontal disease
* Cracked tooth
* Traumatized tooth
* Haemostasis not achieved within 10 minutes

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in radiographic apical status | 3 years
  Change from Baseline Radiographic appearance of apical tissue at 6 months, 1 year, 2 years and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Yu, PhD, Principal Investigator — NUHS

IPD SHARING:
Plan to Share IPD: No